CLINICAL TRIAL: NCT02221024
Title: Randomized Controlled Trial to Evaluate the Efficacy of Normal Saline Flushes at 12 and 24 Hours Intervals in Maintaining Peripheral Intravenous Catheters Patency
Brief Title: Normal Saline Flushes at 12 vs 24 Hours Intervals for Maintaining Peripheral Intravenous Catheters Patency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Ronfani Luca, MD, PhD, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC 10/11
Record Dates: First submitted 2014-08-12; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Pain
Keywords: Peripheral intravenous catheter; Peripheral intravenous lock; Normal saline; Patency; Management; of peripheral; intravenous catheter
MeSH Terms: conditions — Pain | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flushing every 24 hours (Experimental): Flushing with positive pressure with normal saline every 24 hours
  Interventions: Procedure: Flushing with positive pressure; Drug: Normal saline; Device: MicroClave ICU Medica
- Flushing every 12 hours (Active Comparator): Flushing with positive pressure with normal saline every 12 hours
  Interventions: Procedure: Flushing with positive pressure; Drug: Normal saline; Device: MicroClave ICU Medica

INTERVENTIONS:
Procedure: Flushing with positive pressure — Placement of a sterile plug (MicroClave ICU Medica, a neutral displacement connector) on the needle cannula and flushing with positive pressure with saline solution (BD PosiFlush XS Syringes, filled with 3 ml of saline)
Drug: Normal saline
  Other Names: Isotonic saline solution; Physiological saline solution
Device: MicroClave ICU Medica

SUMMARY:
Children admitted in a ward often require a peripheral intravenous catheter to provide access for administration of medications, nutrients, fluids, blood products. Vascular access in children is a frequent and stressful procedure that should be performed as infrequently as possible in order to reduce the child's pain experience and the child's and family's level of distress. The maintenance of patency of indwelling catheters is therefore relevant to minimize need for replacement and children discomfort.

Recent studies investigated the most effective and safe method of maintaining peripheral intravenous lock (peripheral IVL) in children. Most of these studies focused primary on the use of heparin versus saline flushes, showing similar efficacy of the two approaches.

To the best of the investigators knowledge no study addressed the issue of the optimal flushing frequency of normal saline . The aim of this study was to evaluate the efficacy of normal saline flushes, at 12 and 24 hours intervals.

ELIGIBILITY:
Inclusion Criteria:

* age between 1 and 17 years
* peripheral intravenous catheter 22 G or 24 G
* need to maintain the access for at least 24 hours without infusion

Exclusion Criteria:

* need for continuous infusion therapy
* programmed therapy

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2011-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with peripheral intravenous catheter patency | Until catheter use (i.e. drug infusion) or removal (catether related complication or no further need of use), with an expected avarage of 48 hours
  Patency was defined as the possibility of flushing the cannula with a 3 ml Becton Dickinson syringe filled with 3 ml of normal saline in less than 20 seconds without resistance at infusion, pain or erythema

SECONDARY OUTCOMES:
Number of participants with blood extravasation | Until catheter use (i.e. drug infusion) or removal (catether related complication or no further need of use), with an expected avarage of 48 hours
  Presence of blood extravasation in the site of catheter insertion, defined as the presence of changes in the site's appearence and temperature (i.e. edema, blanching, coolness) at the time of nurse's evaluation
Number of participants with pain | Until catheter use (i.e. drug infusion) or removal (catether related complication or no further need of use), with an expected avarage of 48 hours
  Any pain at the site of catheter insertion referred by patients to nurses
Number of participants with skin redness | Until catheter use (i.e. drug infusion) or removal (catether related complication or no further need of use), with an expected avarage of 48 hours
  Presence of skin redness at the site of catheter insertion at the time of nurse's evaluation
Number of participants with swelling | Until catheter use (i.e. drug infusion) or removal (catether related complication or no further need of use), with an expected avarage of 48 hours
  Presence of swelling in the site of catheter insertion at the time of nurse's evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Egidio Barbi, MD, Study Chair — IRCCS Burlo Garofolo, Trieste, Italy; Silvana Schreiber, RN, Study Director — IRCCS Burlo Garofolo, Trieste, Italy
Locations (1):
- Emergency Department, IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia, Italy

REFERENCES:
- [Derived] Schreiber S, Zanchi C, Ronfani L, Delise A, Corbelli A, Bortoluzzi R, Taddio A, Barbi E. Normal saline flushes performed once daily maintain peripheral intravenous catheter patency: a randomised controlled trial. Arch Dis Child. 2015 Jul;100(7):700-3. doi: 10.1136/archdischild-2014-307478. Epub 2015 Jan 14. PMID 25589559